CLINICAL TRIAL: NCT04427345
Title: Predictive Clinical Response Factors in COVID-19 Patients
Brief Title: Predictive Factors COVID-19 Patients
Acronym: MI-COVID
Status: Withdrawn | Type: Observational
Why Stopped: This study has been included in another trial within the same Sponsor
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: MI-COVID
Record Dates: First submitted 2020-06-04; First posted 2020-06-11 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: covid19
Keywords: Coronavirus; sars-covid-2; coronavirus infection
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Covid19 infection related patients: Patients admitted to COVID wards of the S. Gerardo Hospital of Monza, including Intensive Care wards.
  Interventions: Other: Predictive factors for clinical response in patients with COVID-19.

INTERVENTIONS:
Other: Predictive factors for clinical response in patients with COVID-19. — Identify the risk factors for intra-hospital mortality in patients hospitalized in the COVID + hospital wards of the San Gerardo hospital and build a prognostic score through which it is possible to define a stratification that immediately guides the therapeutic choices and the intensity of care .

SUMMARY:
This is a monocentric retro-prospective observational study that will be conducted on all COVID19 positive patients hospitalized at the S. Gerardo Hospital in Monza.

DETAILED DESCRIPTION:
BACKGROUND:

The Severe Acute Respiratory Syndrome-Coronavirus-2 (SARS-CoV-2) pandemic is severely testing the health systems of the most advanced countries. Clinicians are faced with a new pathology of an emerging virus. There is therefore an urgent need to collect real-time clinical data that informs about outcome predictive variables. Furthermore, there are currently no antiviral drugs approved for the treatment of SARS-CoV-2 infection, off-label therapies are being used with drugs already in use for other pathologies that have shown some efficacy in vitro, and some treatments obtained for compassionate use with other drugs that are being tested.

It is more than ever necessary to collect clinical practice data both retrospectively on the work done so far, and in a longitudinal perspective, and analyze them quickly to optimize current treatments and define protocols for the future. Having a good clinical data base also offers the possibility of collaborating with numerous international networks on translational research, which aims to correlate clinical data with virological and immunological data, aimed at the rapid identification of possible specific viral virulence factors, or particular immune structures of the guests who once again define the final clinical outcome.

STUDY DESIGN:

All COVID19 positive patients admitted to San Gerardo Hospital will be enrolled in the study.

After patient signs the informed consent, the following data will be collected:

* birth data
* sex
* demographic data
* comorbidity
* blood chemistry data at the entrance

A series of variables will then be collected relating to the treatment procedure, the therapies, the team's choice to maximize the care ceiling in the individual patient and the entire clinical study of the patient.

STATISTICAL ANALISYS:

Central tendency and dispersion measurements will be used for descriptive analysis of continuous variables while absolute and relative frequencies will be used to describe categorical variables.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years old or above
* Diagnosis of SARS-CoV-2 pneumonia

Exclusion Criteria:

* Explicit refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study involves patients admitted to San Gerardo Hospital from March 1, 2020 to May 31, 2020. The minimum expected follow-up will be one year for all patients.
  Given the nature of the study, no formal calculation of the sample size was made, nor was a sample size predefined. However, given the recruiting potential of the center which in March saw on average 30-60 hospitalizations due to SARS-CoV-2 per day, even considering a progressive decrease in access, it is assumed that the proportion of patients who will be included in the study will exceed 1000 units.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2022-05-12 (Actual)

PRIMARY OUTCOMES:
Identify risk factors for intra-hospital mortality. | Until patient discharge from the hospital (approximately 1 year)
  Identify risk factors for intra-hospital mortality in patients admitted to the COVID + hospital wards of San Gerardo hospital.
Identify risk factors to build a prognostic score. | Until patient discharge from the hospital (approximately 1 year)
  Identify the risk factors to build a prognostic score through which it is possible to define a stratification that immediately guides the therapeutic choices.
Identify risk factors to build a prognostic score. | Until patient discharge from the hospital (approximately 1 year)
  Identify the risk factors to build a prognostic score through which it is possible to define a stratification that immediately directs towards the right intensity of care.

SECONDARY OUTCOMES:
Predictive factors for the hospitalization duration. | Until patient discharge from the hospital (approximately 1 year)
  Description of the predictive factors for the hospitalization duration.
Predictive factors for clinical status patients based on "Ordinal Scale for Clinical Improvement" | Until patient discharge from the hospital (approximately 1 year)
  Description of the predictive factors for the clinical status of patients based on "Ordinal Scale for Clinical Improvement" defined by OMS (
Describe the anti-viral therapies used commonly in this emergency in terms of efficacy | Until patient discharge from the hospital (approximately 1 year).
  Description of efficacy of the anti-viral therapies used today without particular restrictions, but on which solid clinical functioning tests are lacking.
Describe the anti-viral therapies used commonly used in this emergency in terms of safety | Until patient discharge from the hospital (approximately 1 year).
  Description of safety of the anti-viral therapies used today without particular restrictions, but on which solid clinical functioning tests are lacking.
Monitor the clinical course of the disease in discharged patients. | 12 month after discharge
  Description of the disease clinical course in patients 12 months after discharge (mortality, neurological, respiratory and cardiac outcomes).

CONTACTS AND LOCATIONS:
Locations (1):
- ASST Monza-Ospedale San Gerardo, Monza, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosenbaum L. Facing Covid-19 in Italy - Ethics, Logistics, and Therapeutics on the Epidemic's Front Line. N Engl J Med. 2020 May 14;382(20):1873-1875. doi: 10.1056/NEJMp2005492. Epub 2020 Mar 18. No abstract available. PMID 32187459
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Wu C, Chen X, Cai Y, Xia J, Zhou X, Xu S, Huang H, Zhang L, Zhou X, Du C, Zhang Y, Song J, Wang S, Chao Y, Yang Z, Xu J, Zhou X, Chen D, Xiong W, Xu L, Zhou F, Jiang J, Bai C, Zheng J, Song Y. Risk Factors Associated With Acute Respiratory Distress Syndrome and Death in Patients With Coronavirus Disease 2019 Pneumonia in Wuhan, China. JAMA Intern Med. 2020 Jul 1;180(7):934-943. doi: 10.1001/jamainternmed.2020.0994. PMID 32167524
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013